CLINICAL TRIAL: NCT06844201
Title: Postoperative Delirium After Intraoperative Ephedrine Versus Norepinephrine: a Retrospective TriNetX Database Study
Brief Title: Postoperative Delirium After Intraoperative Ephedrine Versus Norepinephrine
Status: Not yet recruiting | Type: Observational
Sponsor: Riverside University Health System Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Baker, Research Coordinator, Riverside University Health System Medical Center
Other Study IDs: Ephedrine vs Norepinephrine
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Ephedrine; Norepinephrine; Postoperative Delirium (POD)
Keywords: Ephedrine; Norepinephrine; Postoperative delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Ephedrine; Norepinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ephedrine group: This group received ephedrine on the day of surgery.
  Interventions: Drug: Ephedrine
- Norepinephrine group: This group received norepinephrine on the day of surgery.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Ephedrine — Received ephedrine the same day of surgery.
  Groups: Ephedrine group
Drug: Norepinephrine — Received norepinephrine the same day of surgery.
  Groups: Norepinephrine group

SUMMARY:
This retrospective study aims to investigate the effects of norepinephrine compared to ephedrine, administered on the day of surgery, on the incidence of postoperative delirium.

DETAILED DESCRIPTION:
This retrospective analysis will be conducted using data from the TriNetX US Collaborative Network. This study was designed to assess the impact of intraoperative norepinephrine versus intraoperative ephedrine use on postoperative delirium. Inclusion criteria includes patients who underwent surgery (CPT code 1003143) and were either administered ephedrine or norepinephrine on the day of surgery and did not receive both vasopressors on the day of surgery. Exclusion criteria exclude patients who underwent neurology and neuromuscular surgery, cardiac surgery, and cardiac procedures; patients who were administered epinephrine or dopamine on the day of surgery; patients who were administered ephedrine or norepinephrine at any time within the 7 days following the day of surgery to account for patients that might have required pressor infusions for other causes; or a prior history of disorientation (ICD-10 code R41.0) or unspecified dementia (F03).

Propensity score matching through TriNetX will be used to adjust for age, sex, race, BMI, and comorbidities including cerebrovascular disease (ICD-10 code I60-I69), chronic heart failure (I11.0), primary hypertension (I10, I11.9), chronic obstructive pulmonary disease (COPD) (J42, J43, J44, J47), asthma (J45), chronic kidney disease (CKD) (I12, I13), diabetes mellitus (E08-E13), depression (F32.A), schizoaffective disorders (F25), alcohol and drug abuse (F10.1, F10.2, Z71.4), smoking status (F17.2, F17.21), and history of antipsychotic (CN700) and benzodiazepine (C302) usage.

Independent t-tests and chi-squared tests will be used to compare postoperative delirium across the cohorts. To evaluate the relationship between norepinephrine and postoperative delirium versus ephedrine and postoperative delirium, risk differences, and risk ratios with 95% CIs will be calculated following propensity score matching. The TriNetX platform will be used for all analyses, with p < 0.05 representing statistical significance.

ELIGIBILITY:
Ephedrine group:

Inclusion Criteria:

* underwent surgery (CPT code 1003143)
* administered ephedrine on the day of surgery

Exclusion Criteria:

* received both vasopressors (ephedrine and norepinephrine) on the day of surgery.
* patients who underwent neurology and neuromuscular surgery, cardiac surgery, and cardiac procedures
* patients who were administered epinephrine or dopamine on the day of surgery
* patients who were administered ephedrine or norepinephrine at any time within the 7 days following the day of surgery
* a prior history of disorientation (ICD-10 code R41.0) or unspecified dementia (F03)

Norepinephrine group:

Inclusion Criteria:

* underwent surgery (CPT code 1003143)
* administered norepinephrine on the day of surgery

Exclusion Criteria:

* received both vasopressors (ephedrine and norepinephrine) on the day of surgery.
* patients who underwent neurology and neuromuscular surgery, cardiac surgery, and cardiac procedures
* patients who were administered epinephrine or dopamine on the day of surgery
* patients who were administered ephedrine or norepinephrine at any time within the 7 days following the day of surgery
* a prior history of disorientation (ICD-10 code R41.0) or unspecified dementia (F03)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients within the TriNetX database.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | Within 7 days following surgery.
  The outcome of postoperative delirium will be observed using the ICD-10 codes F05, R40, and R41 for delirium, somnolence, and disorientation, respectively.

IPD SHARING:
Plan to Share IPD: No
We do not have an IPD in place at this time.